CLINICAL TRIAL: NCT00620945
Title: Use of Phenoxybenzamine [PBZ] IV to Assist High Flow Low Pressure Perfusion [HFLPP] on Cardio-pulmonary Bypass in Infants and Children With Congenital Heart Disease and to Assist Steady State Alfa-blockade in the Intensive Care Phase
Brief Title: Use of Phenoxybenzamine [PBZ] IV to Assist High Flow Low Pressure Perfusion [HFLPP] on Cardio-pulmonary Bypass
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New protocol now being used for cardiopulmonary bypass
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCF IRB # 06-494
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Congenital Heart Surgery; Cardiopulmonary Bypass
Keywords: Congenital heart surgery; Cardiopulmonary bypass; Phenoxybenzamine
MeSH Terms: interventions — Phenoxybenzamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Treatment Group
  Interventions: Drug: Phenoxybenzamine

INTERVENTIONS:
Drug: Phenoxybenzamine — Use of Phenoxybenzamine:
  Loading dose given at the time of going on CPB:
  * For patients with obstructing lesions on systemic side:
    * 0.25 mg/kg dose in the bypass circuit
    * None intravenous
  * For patients without obstructing left sided lesions:
    * 0.5 mg/kg in the bypass circuit
    * 0.5 mg/kg I.V. at cannulation
  Maintenance dose given in the post-operative period:
  * 0.3 mg/kg I.V. every 8 hours till oral intake is started or for first 48 hours
  * 0.3 mg/kg P.O. every 8 hours for next 24 hours
  * 0.15 mg/kg P.O. every 8 hours for next 24 hours and then stop
  * Hold PBZ if the patient is on norepinephrine infusion or the mean arterial pressure is lower than that allowed for the age group
  Other Names: Dibenzyline

SUMMARY:
Cardiopulmonary bypass [CPB] in small size bodies can result in decreased peripheral perfusion. This results in anaerobic metabolism as evidenced by lactic acidosis. High flow perfusion results in systemic hypertension which is accentuated by moderate hypothermia commonly used during cardiopulmonary bypass. Phenoxybenzamine [PBZ] is an arteriolar vasodilator that acts by irreversibly blocking the alpha adrenergic receptors. It causes vasodilatation allowing high flow, low pressure CPB. It has been used extensively outside US in Canada, Europe and Australia. In the US oral PBZ is FDA approved, whereas intravenous PBZ is only available as an investigational drug

DETAILED DESCRIPTION:
Background Cardiopulmonary bypass [CPB] in small size bodies can result in decreased peripheral perfusion. This results in anaerobic metabolism as evidenced by lactic acidosis. High flow results in systemic hypertension which is accentuated by moderate hypothermia commonly used during cardiopulmonary bypass. Phenoxybenzamine [PBZ] is an arteriolar vasodilator that acts by irreversibly blocking the alpha adrenergic receptors. It causes vasodilatation allowing high flow, low pressure CPB. It has been used extensively outside US in Canada, Europe and Australia. In the US oral PBZ is FDA approved, whereas intravenous PBZ is only available as an investigational drug. At the Cleveland Clinic this medication has been used under this protocol since 1994 in >1000 without any significant or serious adverse outcome. The drug is also used at Texas Children's Hospital, Hospital for Sick Children in Toronto, Children's Hospital of Wisconsin and a number of centers throughout Europe, Australia and Asia. The drug has helped reduce the mortality of children undergoing cardiopulmonary bypass.

The theoretic benefit of PBZ in this patient population is uniform and smooth reduction fo systemic vascular resistance in the perioperative period. This uniform systemic vasodilation allows low pressure, high flow systemic perfusion on cardiopulmonary bypass. We feel that this ins in part responsible for improved outcome after cardiopulmonary bypass, including less end-organ edema formation and dysfunction. Due to experience in this and other centers we strongly believe that the use of PBZ in the bypass management protocol of these patients represents the state-of-the-art and not an experimental investigation. Since in the US the drug is not available except as an investigational drug, we have been required to use it as an investigational new drug [IND] PBZ[oral] is currently used in the US for the management of pheochromocytoma. It has a proven track record and known to be safe. Use in a large number of patients worldwide has shown no serious side-effects except hypotension [which is an effect indeed] requiring norepinephrine [an alpha agonist commonly used after cardiopulmonary bypass in these patients anyway].

Patients

The following patients are candidates for receiving PBZ for HFLPP. These include:

1. All patients under 16 kg.
2. Those patients between 16-18 kg whose pre bypass hemoglobin is <16 g/dl
3. All patients are less than 18 years of age.

Use of Phenoxybenzamine:

Loading dose given at the time of going on CPB:

* For patients with obstructing lesions on systemic side:

  * 0.25 mg/kg dose in the bypass circuit
  * None intravenous
* For patients without obstructing left sided lesions:

  * 0.5 mg/kg in the bypass circuit
  * 0.5 mg/kg I.V. at cannulation

Maintenance dose given in the post-operative period:

* 0.3 mg/kg I.V. every 8 hours till oral intake is started or for first 48 hours
* 0.3 mg/kg P.O. every 8 hours for next 24 hours
* 0.15 mg/kg P.O. every 8 hours for next 24 hours and then stop
* Hold PBZ if the patient is on norepinephrine infusion or the mean arterial pressure is lower than that allowed for the age group
* Do not use maintenance dose in the following patients unless they are on maximum dose of sodium nitroprusside infusion and still hypertensive:

  * Norwood patients
  * Fontan patients
  * Patients with residual left ventricular obstructive lesions - don't use at all in the post operative period

Data collected and monitored for the purpose of this study only:

Demographic information, side effects and mortality data would be recorded and kept in a password protected computer in a secure-access-only physician office. Only composite data without individual identifiers will be reported to the IRB and FDA. No publication is planned from this study and no follow-up will be done after the patient is discharged from the hospital.

Side effects to be monitored:

* Hypotension requiring norepinephrine in excess of usual dose [0.2 micrograms/kg/min]
* Death from such hypotension in the absence of other causes [such as bleeding, sepsis]
* Effects occuring within 12 hours of I.V. dose administration or within 24 hours of P.O. dose administration
* Any unanticipated or unusual side effects [none noted since 1994] Consent Informed consent would be obtained from the parents/guardians of all patients. Assent will be obtained from children of >7 years age.

ELIGIBILITY:
Inclusion Criteria:

Patients

The following patients are candidates for receiving PBZ for HFLPP. These include:

1. All patients under 16 kg.
2. Those patients between 16-18 kg whose pre bypass hemoglobin is <16 g/dl
3. All patients are less than 18 years of age

Exclusion Criteria:

1. Those with bloodless prime in Cardiopulmonary bypass circuit
2. Age > 18years
3. Wt. >16 kg

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 87 (Actual)
Dates: Start 2006-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad A Mumtaz, MD, Principal Investigator — The Cleveland Clinic

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of Recruitment: June 2006 to September 2008
Groups:
- Phenoxybenzamine Treatment: Treatment Group- patients treated with phenoxybenzamine
Period: Overall Study
Arm/Group | Phenoxybenzamine Treatment
Started | 87 (Total number in the study)
Completed | 87
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients undergoing open heart surgery and who are less than 18 years of age.
Groups:
- Phenoxybenzamine: Treatment Group
  Phenoxybenzamine: Use of Phenoxybenzamine:
  Loading dose given at the time of going on CPB:
  * For patients with obstructing lesions on systemic side:
    * 0.25 mg/kg dose in the bypass circuit
    * None intravenous
  * For patients without obstructing left sided lesions:
    * 0.5 mg/kg in the bypass circuit
    * 0.5 mg/kg I.V. at cannulation
  Maintenance dose given in the post-operative period:
  * 0.3 mg/kg I.V. every 8 hours till oral intake is started or for first 48 hours
  * 0.3 mg/kg P.O. every 8 hours for next 24 hours
  * 0.15 mg/kg P.O. every 8 hours for next 24 hours and then stop
  * Hold PBZ if the patient is on norepinephrine infusion or the mean arterial pressure is lower than that allowed for the age group
Arm/Group | Phenoxybenzamine
Number analyzed (Participants) | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 87
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 87

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving High Flow Low Pressure on Cardiopulmonary Bypass
Description: Percentage of patients who achieved high flow, low pressure on cardiopulmonary bypass
Time Frame: From time of cardiopulmonary bypass initiation until the time that high flow, low pressure on cardiopulmonary bypass was achieved, assessed up to 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Phenoxybenzamine Treatment
Number analyzed (Participants) | 87
Participants | 87

2. Secondary Outcome: Mortality
Description: Percentage of patients who died within 30 days of the procedure
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phenoxybenzamine Treatment
Number analyzed (Participants) | 87
Participants | 5

ADVERSE EVENTS:
Arm/Group | Phenoxybenzamine
All-Cause Mortality (participants affected / at risk) | 5/87
Serious Adverse Events (participants affected / at risk) | 5/87
Other Adverse Events (participants affected / at risk) | 0/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenoxybenzamine (N=87)
Myocardial dysfunction (Cardiac disorders) | 3 (3) — Cause of death was myocardial dysfunction, pulmonary hypertension, or myocardial infarction
Pulmonary hypertension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Due to a change in leadership the protocol of cardiopulmonary bypass was changed on 9/22/2008. The high flow low pressure perfusion is no longer used. As a result phenoxybenzamine was no longer able to be studied and the study was closed early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No